CLINICAL TRIAL: NCT00626171
Title: A Study Evaluating the Role of Cigarette Smoking in Regulating Allergen-induced Early and Late Responses in Mild Asthmatics.
Brief Title: Role of Cigarette Smoking in Regulating Allergen-induced Early and Late Responses in Mild Asthmatics
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Paul O'Byrne, Paul O'Byrne, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ZMsmsp
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Asthma
Keywords: smoking; asthma; sputum
MeSH Terms: conditions — Asthma; Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Allergen challenge
  Interventions: Procedure: Allergen Challenge

INTERVENTIONS:
Procedure: Allergen Challenge — Allergen challenge

SUMMARY:
The objective of this study is to determine the effect of cigarette smoking on inflammatory cell recruitment to the lungs after an allergen challenge, in non-smoking and currently smoking mild asthmatic subjects.

When comparing non-smoking asthmatics to smoking asthmatics, do differential cell counts obtained from inflammatory cells in induced sputum after allergen challenge differ?

Will differential cell counts show a decline in inflammatory cells in the induced sputum of asthmatics who have refrained from smoking for eight weeks?

This study is a randomized, case-controlled study. The first part of the study requires smoking and non-smoking subjects who will attend 2 study periods of 3 consecutive days (triad). In each triad, they will be challenged with allergen or diluent by inhalation, in a random order, and each triad is separated by a washout period. In the second part of the study, current smokers will be invited to undergo another allergen challenge 8 weeks of smoking cessation.

DETAILED DESCRIPTION:
10 non-smoking adult subjects and 10 smoking adult subjects with mild atopic asthma will be studied.

Part 1: On the first study day of the triad, subjects will undergo screening procedures, including complete history and physical examination. Methacholine inhalation challenge and allergen skin titration will be performed to determine the concentration of allergen required for inhalation. Sputum will be induced for baseline measurement of airway inflammatory cells. On the second day, subjects will inhale the allergen or diluent in randomized order, and spirometry will be measured for the next 7 hours. Sputum will be collected at 7 hours after challenge. On the third day, subjects will report to the lab 24 hours after allergen/diluent inhalation challenge. Sputum cells will be collected to measure the percentage of airway inflammatory cells, including eosinophils and neutrophils. After washout of 2-4 weeks, subjects will return to undergo diluent/allergen triad.

Part 2: Asthmatic smokers will be studied to investigate allergen-induced changes in inflammatory cell numbers after they quit smoking for a period of 8 weeks. Asthmatic smokers who were involved in the first part of the study will be asked if they would like to participate in this part of the study, and they will be provided with smoking cessation tools including nicorette gum and nicotine patches, to aid them in ceasing to smoke. At the beginning of the study period, the same procedures that occurred in part 1 will be performed to obtain initial baseline results- ie- history, physical examination, skin prick test, methacholine challenge and sputum induction. Throughout the 8 week period, subjects will be required to come in weekly to perform a carboxyhemoglobin test, to ensure that they have not been smoking that week. At the end of the 8 week period, an allergen challenge triad will be carried out (as was performed in Part 1 of the study). Those subjects who were not able to comply to the smoking cessation regime will still be included in the final measurements.

We hypothesize that inflammatory cell counts will be higher in the asthmatic smokers versus asthmatic non-smokers. We also hypothesize that subjects who quit smoking for the 8 week period will show a decline in inflammatory cell counts indicating an improvement in lung function.

We believe that the results of this novel study will provide greater insight into the inflammatory response in asthmatic smokers, and will suggest appropriate therapeutic approaches for control of asthma in smokers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with mild atopic asthma, presently well controlled on ß2-agonist only.
* Baseline FEV1 more than or equal to 70% of predicted normal.

Exclusion Criteria:

* Past or present cardiovascular, renal, liver or endocrine disease.
* Airway infection during the last 4 weeks.
* Exacerbation during the last 4 weeks.
* Inhaled or oral steroids during the last 4 weeks.
* Anti-asthma medication other than inhaled and/or oral ß2-agonists during the last 4 weeks.
* Pregnant or lactating women or women actively seeking pregnancy or lack of adequate contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To measure the number of inflammatory cells in induced sputum following allergen challenge in smoking and non-smoking asthmatic subjects. | 7h and 24 h post

CONTACTS AND LOCATIONS:
Overall Officials: Paul O'Byrne, MD, Principal Investigator — McMaster University; Gail Gauvreau, PhD, Study Director — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada